CLINICAL TRIAL: NCT04925323
Title: VALIDATION OF A GMP-COMPLIANT BIOPRINTING PROCESS FOR MANUFACTURING A DERMO-EPIDERMAL AUTOLOGOUS SKIN SUBSTITUTE FOR FURTHER THERAPEUTIC USE
Brief Title: A DERMO-EPIDERMAL AUTOLOGOUS SKIN SUBSTITUTE FOR FURTHER THERAPEUTIC USE
Acronym: BIOPSKIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-33; 2020-A01599-30 (Other: IDRCB)
Record Dates: First submitted 2021-03-29; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Plastic Surgeries
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a plastic or repair surgery indication generating surgical waste (Experimental)
  Interventions: Biological: BLOOD SAMPLES; Biological: surgical tissue samples

INTERVENTIONS:
Biological: BLOOD SAMPLES — BLOOD SAMPLES
Biological: surgical tissue samples — unused surgical tissue removed during plastic surgeries

SUMMARY:
Innovative technologies in the emerging field of regenerative medicine might allow an improvement in the treatment of deep complex wounds leading to faster and better wound healing. Among them, the bioprinting technology, consisting in "printing human cells and biomaterials" to create a "dermo-epidermal substitute" that mimics an alternative of the physiological skin is the most promising alternative.

Besides improving skin substitutes properties, bioprinting allows to translate the manufacturing process of tissue-engineered products from manual, operator-dependent processes to a reproducible and automated solution. This paves the way to the manufacturing of therapeutic bioprinted products at the point of care, as close as possible from patients.

DETAILED DESCRIPTION:
In this preclinical in vitro study, the investigators plan to generate GMP-compliant validation batches of "bio-printed dermo-epidermal substitutes" from 25 healthy volunteer patients' unused surgical tissue removed during plastic surgeries.

Volunteer's harvested tissue will allow to extract and then amplify the epidermal keratinocytes and dermal fibroblasts. Successive cultures and bioprinting steps will generate a "bio-printed dermo-epidermal substitute" in 2 or 3 weeks. A blood test may also be performed on the volunteers to characterize the genetic stability during the different stages of the process.

ELIGIBILITY:
Inclusion Criteria:

* Adult adult males or females
* Members of a social security scheme.
* No contraindications to general anesthesia
* Relevant to a plastic or repair surgery indication generating surgical waste.

Exclusion Criteria:

* Pregnant and/or nursing women
* Persons deprived of liberty
* Major under guardianship
* Persons unable to read the backgrounder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
bioprinted dermo epidermal substitute sterility assessment | 24 MONTHS
  Culture media from dermo-epidermal bioprinted substitutes were sampled in Bactec culture bottles (Peds Plus Aerobic/F and Plus Anaerobic/F culture vials, containing each 40 mL of medium). The Bactec method (Becton Dickinson, Sparks, MD, USA) uses a computer-controlled incubation/detection system. The media used contained proprietary factors designed to inactivate a wide variety of antibacterial and antifungal agents. Bactec culture bottles were incubated at 37 °C for a total of 10 days, and automated readings were taken every 10 min. Detection of organisms resulted in an audible alarm and automatic recording of time to detection.
Population Doubling Rate of keratinocytes | 24 MONTHS
Population Doubling Rate of fibroblasts | 24MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — AP HM; Dominique CASANOVA, Principal Investigator — AP HM
Locations (1):
- assistance publique hôpitaux de Marseille, Marseille, France